CLINICAL TRIAL: NCT04933318
Title: Effects of TENS and Interference on Pain, Functional Status and Range of Motion in Shoulder Pain in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Yeşil (Other)
Responsible Party: Sponsor-Investigator, Hilal Yeşil, Assoc.Prof., Afyonkarahisar Health Sciences University
Organization: Afyonkarahisar Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYSHHO
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Hemiplegic Shoulder Pain
Keywords: Rehabilitation; Exercise; TENS
MeSH Terms: conditions — Motor Activity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcutaneous electrical nerve stimulation (TENS) (Active Comparator): Transcutaneous electrical nerve stimulation (TENS)- analgesic current therapy
  Interventions: Other: TENS
- shamTENS (Sham Comparator): shamTranscutaneous electrical nerve stimulation (TENS)- analgesic current therapy
  Interventions: Other: shamTENS
- Interferential current therapy (IFC) (Active Comparator): Interferential current therapy (IFC)- analgesic current therapy
  Interventions: Other: IFC
- shamIFC (Sham Comparator): shamInterferential current therapy (IFC)- analgesic current therapy
  Interventions: Other: shamIFC

INTERVENTIONS:
Other: TENS — Transcutaneus electrical nerve stimulation (TENS)- analgesic current therapy
  Arms: Transcutaneous electrical nerve stimulation (TENS)
Other: shamTENS — shamTranscutaneus electrical nerve stimulation (shamTENS)- analgesic current therapy
  Arms: shamTENS
Other: IFC — Interferential current therapy (IFC)- analgesic current therapy
  Arms: Interferential current therapy (IFC)
Other: shamIFC — shamInterferential current therapy (shamIFC)- analgesic current therapy
  Arms: shamIFC

SUMMARY:
Effects of TENS and Interference on Pain, Functional Status and Range of Motion in Shoulder Pain in Stroke Patients

DETAILED DESCRIPTION:
Hemiplegic shoulder pain treatment methods are, analgesics, local steroid injection, physical therapy modalities and exercise. There are publications about the use of TENS and interferential currents (IFC) in the treatment of hemiplegia related shoulder pain and their effectiveness. However when we look at the literature, we did not find a study that evaluated the efficacy of TENS and IFC in hemiplegic shoulder pain. For this reason, in this study, we aimed to determine the effects of these analgesic treatment modalities on the patient's pain, functional status and shoulder range of motion (ROM) in these patients. 60 stroke patients with shoulder pain randomized to four treatment groups. 15 patients in Group 1 were given TENS treatment to the shoulder area for 25 minutes by conventional method ( 20 sessions, 5 times a week), then, a classical stroke rehabilitation program was applied under the guidance of a physiotherapist.. 15 patients in Group 2 were given shamTENS treatment to the shoulder area for 25 minutes ( 20 sessions, 5 times a week), then, a classical stroke rehabilitation program was applied under the guidance of a physiotherapist.15 patients in Group 3 were given 100 Hz IFC treatment to the shoulder area for 25 minutes ( 20 sessions, 5 times a week), then, a classical stroke rehabilitation program was applied under the guidance of a physiotherapist. 15 patients in Group 4 were given shamIFC treatment to the shoulder area for 25 minutes ( 20 sessions, 5 times a week), then, a classical stroke rehabilitation program was applied under the guidance of a physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

1.Having shoulder pain due to hemiplegia 2- Having had hemiplegia in the last 8 months 3- Having hemiplegia for the first time 4- Not having a problem in the painful shoulder before hemiplegia 5- normal light touch and pinprick tests of the affected shoulder 6- pain level in the affected extremity as measured by VAS is at least 4 7- Brunnstrom upper extremity stage with 1-2-3

Exclusion Criteria:

1. Neoplasia
2. uncontrolled hypertension
3. Serious arrhythmias
4. Having pacemakers
5. Epilepsy
6. Severe sensory impairment, wound, infection in the application area
7. bleeding disorders

9. Uncooperative patients 10- Patients with acute infection 11- Patients with a history of trauma to the painful shoulder 12- Treatment for pain in the affected shoulder (blockage, intra-articular injection, and physical therapy agent)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline VAS (visual analog scale) at 4th and 8th week | up to 8 weeks
  The patients were asked to make an assesment of their pain level between 0 and 10 scale

SECONDARY OUTCOMES:
Change from baseline quality of life (short form 36) at 4th and 8th week | up to 8 weeks
  The physical and mental health summary scores were the primary components used. Scoring is on a scale of 0 to 100 and a higher score reflects better health-related quality of life.
Change from baseline shoulder range of motion (ROM) at 4th and 8th week | up to 8 weeks
  The patients' shoulder joint range of motion will be measured with a goniometer.
Change from baseline Beck depression inventory (BDI) at 4th and 8th week | up to 8 weeks
  A total Beck score (0-63) is obtained by giving each question a score of 0-3 in the survey. 17 is considered the threshold value for the degree of depression.
Change from baseline Brunnstrom staging at 4th and 8th week | up to 8 weeks
  According to Brunnstrom, the motor recovery of the hemiplegic patient is divided into six stages. These stages are defined according to muscle tone and extremity synergies. Stage 1: The involved side is flaccid, there is no active movement. Stage 6: Isolated joint movement is freely available.
Change from baseline Functional ambulation score (FAS) at 4th and 8th week | up to 8 weeks
  It is used to evaluate the support patients need during walking. It has 5 phases. STAGE 0: Non-functional ambulation: The patient does not walk, he can only walk on the parallel bar. STAGE 5: There is independent ambulation.
Change from baseline functional independence measure (FIM) at 4th and 8th week | up to 8 weeks
  FIM consists of 2 parts: motor and cognitive skills. Each of the sections contains 18 sub-items under 6 main items (self-care, sphincter control, mobility and transfer, mobility and walking, communication and social perception). The lowest score that can be obtained from the scale is 18, and the highest score is 126.
Change from baseline modified ashworth scale (MAS) at 4th and 8th week | up to 8 weeks
  It is used when evaluating the upper extremity muscle tone of patients. Stages on this scale: 0: Muscle tone is normal. 4: The affected parts are rigid in flexion and extension, there is a severe increase in tone.
Change from baseline fugl meyer assessment at 4th and 8th week | up to 8 weeks
  It is a stroke-specific, performance-based scale, with each parameter being 0; fail, 1; partially successful and 2; is scored as a completely successful performance. It is based on the motor recovery stages of Twitchell and Brunnstrom.
Change from baseline Shoulder Disability Questionnaire (SDQ) at 4th and 8th week | up to 8 weeks
  It is a 16-item pain-related disability questionnaire describing common conditions that exacerbate symptoms in patients with shoulder disease. A score of zero indicates maximum well-being, and a score of 100 indicates maximum ill health.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Yesil, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Hilal Yeşil, Merkez, Afyonkarahisar, Turkey (Türkiye)